CLINICAL TRIAL: NCT07164131
Title: Azithromycin Versus Doxycycline in Hospitalized Adult Patients With Community Acquired Pneumonia Treated With Beta-lactams
Acronym: AD-CAP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Yewande Odeyemi, MD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-006503
Record Dates: First submitted 2025-08-20; First posted 2025-09-09 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Community-acquired Pneumonia
Keywords: Azithromycin; Doxycycline; hospitalized
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Doxycycline; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Doxycycline group (Active Comparator): Subjects hospitalized for community acquired pneumonia will receive standard of care treatment with Doxycycline
  Interventions: Drug: Doxycycline
- Azithromycin group (Active Comparator): Subjects hospitalized for community acquired pneumonia will receive standard of care treatment with Azithromycin
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Doxycycline — Subjects will receive Doxycycline (orally or intravenously) in combination with beta-lactam therapy within 12 hours of hospital admission. Treatment duration will be 5-7 days.
  Arms: Doxycycline group
Drug: Azithromycin — Subjects will receive Azithromycin (orally or intravenously) in combination with beta-lactam therapy within 12 hours of hospital admission. Treatment duration will be 5-7 days.
  Arms: Azithromycin group

SUMMARY:
The purpose of this study is to compare effectiveness and safety of Azithromycin versus Doxycycline in adult patients hospitalized with community acquired pneumonia (CAP) treated with Beta-lactams.

ELIGIBILITY:
Inclusion Criteria:

• All adult patients (>18 years old) admitted with CAP and receiving a beta-lactam antibiotic plus a form of atypical coverage (azithromycin or doxycycline) in the ED within 12 hours of admission.

Exclusion Criteria:

* High clinical suspicion for Legionella pneumonia
* Allergy or contraindication to the use of either azithromycin or doxycycline (usual clinical practice)
* Antibiotics not for CAP
* Pregnant women (based on clinical assessment as part of standard of care)
* Severe CAP as defined by the ATS/IDSA criteria
* Corrected QT prolongation (> 440 ms in men and > 460 ms in women)
* Receiving a different antibiotic (e.g quinolones)
* Admission > 24 hours
* Known to be a prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1120 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2030-09-01 (Estimated); Study Completion 2031-09-01 (Estimated)

PRIMARY OUTCOMES:
Hospital-free days | 28 days
  Number of days subject remained out of hospital

SECONDARY OUTCOMES:
Oxygen-free days | 28 days
  Number of days subject does not require new supplemental oxygen use. Oxygen-free days will be set as 0 for patients who died during the stay or had a length of stay of ≥28 days
180-day mortality | 180 days
  Defined as mortality at 180 days after discharge
Need for advanced respiratory support or in-hospital mortality | Up to 28 days
  Defined as a composite of need for advanced respiratory support or mortality during hospitalization. Need for advanced respiratory support would include need for high flow nasal cannula, non-invasive positive pressure ventilation, and invasive ventilation in patients not requiring this at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Yewande Odeyemi, Principal Investigator — Mayo Clinic
Locations (5):
- United States (5):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic Health System-Mankato, Mankato, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mayo Clinic Health System-La Crosse, La Crosse, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials